CLINICAL TRIAL: NCT03114371
Title: Effects of Intranasal Administrations of Oxytocin on Behavioural Troubles, Hyperphagia and Social Skills in Children With Prader-Willi Syndrome Aged From 3 to 12 Years.
Brief Title: Oxytocin Intranasal Administrations in Children With Prader-Willi Syndrome Aged From 3 to 12 Years
Acronym: Oxyjeune
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15 7837 03; 2016-003273-18 (EudraCT Number)
Record Dates: First submitted 2017-03-10; First posted 2017-04-14 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Prader-Willi Syndrome
Keywords: Prader-Willi syndrome; Oxytocin; Behavioural troubles
MeSH Terms: conditions — Prader-Willi Syndrome | interventions — Oxytocin

STUDY DESIGN:
Intervention Model Description: Children will receive after randomization either placebo or oxytocin administration (daily intranasal) for a total duration of 12 consecutive weeks.
Who Masked: Participant, Investigator
Masking Description: The packaging, presentation and labelling of the bottles used during the blind phase will guarantee the blindness to the healthcare team and the patient.
  The allocation of the treatment arms to each treatment number will be carried out according to the randomization table established beforehand.
  Until the end of the study, neither the investigating physician nor the patient will know the group to which the patient has been randomly assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxytocin (Experimental): Daily intranasal administrations of oxytocin for 12 weeks, followed by an open-label period of 12 weeks of oxytocin. Oxytocin dose will be 8 International Unit for patients aged from 3 to 6 years and 16 International Unit for patients aged from 7 to 12 years.
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Daily intranasal administrations of placebo for 12 weeks, followed by an open-label period of 12 weeks of oxytocin. Oxytocin dose will be International Unit for patients aged from 3 to 6 years and 16 International Unit for patients aged from 7 to 12 years.
  Interventions: Drug: Placebo; Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin — The study drug is oxytocin in intra-nasal administration, Syntocinon®, reconditioned as a placebo-like spray. The dosage administered will be 8 International Unit, ie 1 spray (4 International Unit per spray) in each nostril per day for the first 12 weeks, in 3 and 6 years old patients. The dosage administered will be 16 International Unit or 2 sprays in each nostril per day for the first 12 weeks, in 3 to 6 years old patients.
  Other Names: Intranasal administration of oxytocin (Week 1 to 12)
  Arms: Oxytocin
Drug: Placebo — Placebo should be used as a spray, similar to that of the oxytocin. The dosage administered will be 1 spray in each nostril per day for the first 12 weeks in 3 to 6 years old patients. The dosage administered will be 2 sprays in each nostril per day for the first 12 weeks, in 7 to 12 years old patients.
  Other Names: Intranasal administration of placebo (Week 1 to 12)
  Arms: Placebo
Drug: Oxytocin — Each patient will receive oxytocin in open label (Syntocinon® not reconditioned) from week 13 to week 24 according to the same dosages.
  Other Names: Intranasal administration of oxytocin (Week 13 to 24)

SUMMARY:
Positive results in preclinical and clinical studies in adults and infants with Prader-Willi syndrome lead investigators to set up a new study in children with Prader-Willi syndrome. The objective of this study is to document effects of oxytocin intranasal administrations on behavioural troubles in children with Prader-Willi syndrome aged from 3 to 12 years.

DETAILED DESCRIPTION:
Two groups of patients will be constituted according to their age; "Group 1" children aged from 3 to 6 years (n = 20) and "Group 2" children aged from 7 to 12 years (n = 20). Within each group, subjects will be randomized to receive either oxytocin or placebo for 12 consecutive weeks. A second period of 12 consecutive oxytocin treatment weeks will then be performed for all patients, followed by a 4-week observation period to document effects after discontinuation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patient with a complete genetic diagnosis of Prader-Willi syndrome
* patient treated by growth hormone for at least 1 year
* patient naïve for oxytocin for at least 5 years

Exclusion Criteria:

* patient who do not accept intranasal administrations (major behavioural trouble)
* patient with hepatic insufficiency : serum transaminases (SGOT, SGPT) higher than 3 times normal values for age
* patient with renal insufficiency : serum creatinine higher than 3 times normal values for age
* patient with an antecedent of abnormal electrocardiogram
* patient with arterial hypertension or hypotension
* patient with type 1 or 2 diabetes

Ages: 3 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2016-11-28 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Evolution of behavioural troubles evaluated by the global score of Child Behavior Check List Questionnaire after 12 weeks of oxytocin/placebo treatment. | Week 12
  It's variation between inclusion and 12 weeks of total score total problems from the Child Behavior Check List Questionnaire.

SECONDARY OUTCOMES:
Evaluation of hyperphagia after 12 weeks of oxytocin/placebo treatment. | Week 12
  It is the variation of each of the three sub-scores obtained from the Dykens hyperphagia questionnaire between day 0 and week 12.
Evaluation of social skills after 12 weeks of oxytocin/placebo treatment. | Week 12
  It is variation between day 0 and week 12 of the total score obtained from the social skills assessment questionnaire for children aged from 3 to 6 years and the Social Responsiveness Scale questionnaire for children aged from 7 to 12 years.
Evaluation of auto- and hetero-aggressive after 12 weeks of oxytocin/placebo treatment. | Week 12
  It is variation between day 0 and week 12 of the total score obtained from the self-aggression assessment questionnaire.
Evaluation of psychopathology after 12 weeks of oxytocin/placebo treatment. | Week 12
  It is the variation of the following sub-scores obtained from the Child Behaviour Check List questionnaire (only the following 3 subscales) between day 0 and week 12.
Evaluation of global clinical status after 12 weeks of oxytocin/placebo treatment. | Weeks 12
  It is improvement of the patient's overall clinical condition after 12 weeks of treatment with oxytocin/placebo. It's assessed by the Clinical Global Impression Scale's score.
  This scale of improvement of Clinical Global Impression is a 7-point ordinal qualitative scale of "very greatly improved" rated + 3 to "very strongly aggravated" rated -3. The result is expressed in total score which varies from -3 to +3.
Evaluation of acyl and desacyl ghrelin plasma levels after 12 weeks of oxytocin/placebo treatment. | Week 12
  It is evolution of circulating levels of acylated and deacylated ghrelin will be the variations of these rates and the variation of the relationships between day 0 and week 12.
Evaluation of attentional abilities after 12 weeks of oxytocin/placebo treatment, for patients aged from 7 to 12 years at inclusion. | Week 12
  It is evolution of attentional abilities is evaluated by a computerized test, the Attention Network Test.
Evaluation of metabolic brain resting state after 12 weeks of oxytocin/placebo treatment, for patients aged from 7 to 12 years at inclusion. | Week 12
  It is evolution of metabolic brain resting state is evaluated by a magnetic resonance imaging to study the cerebral metabolism between day 0 and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Sophie ÇABAL-BERTHOUMIEU, Dr, Principal Investigator — Centre de référence du syndrome de Prader-Willi, Hôpital des Enfants
Locations (1):
- Centre de référence du syndrome de Prader-Willi Hôpital des Enfants, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bittel DC, Kibiryeva N, Sell SM, Strong TV, Butler MG. Whole genome microarray analysis of gene expression in Prader-Willi syndrome. Am J Med Genet A. 2007 Mar 1;143A(5):430-42. doi: 10.1002/ajmg.a.31606. PMID 17236194
- [Background] Constantino JN, Todd RD. Intergenerational transmission of subthreshold autistic traits in the general population. Biol Psychiatry. 2005 Mar 15;57(6):655-60. doi: 10.1016/j.biopsych.2004.12.014. PMID 15780853
- [Background] Dykens EM, Lee E, Roof E. Prader-Willi syndrome and autism spectrum disorders: an evolving story. J Neurodev Disord. 2011 Sep;3(3):225-37. doi: 10.1007/s11689-011-9092-5. Epub 2011 Aug 20. PMID 21858456
- [Background] Dykens EM, Maxwell MA, Pantino E, Kossler R, Roof E. Assessment of hyperphagia in Prader-Willi syndrome. Obesity (Silver Spring). 2007 Jul;15(7):1816-26. doi: 10.1038/oby.2007.216. PMID 17636101
- [Background] Dykens E, Schwenk K, Maxwell M, Myatt B. The Sentence Completion and Three Wishes tasks: windows into the inner lives of people with intellectual disabilities. J Intellect Disabil Res. 2007 Aug;51(Pt 8):588-97. doi: 10.1111/j.1365-2788.2006.00937.x. PMID 17598872
- [Background] Einfeld SL, Smith E, McGregor IS, Steinbeck K, Taffe J, Rice LJ, Horstead SK, Rogers N, Hodge MA, Guastella AJ. A double-blind randomized controlled trial of oxytocin nasal spray in Prader Willi syndrome. Am J Med Genet A. 2014 Sep;164A(9):2232-9. doi: 10.1002/ajmg.a.36653. Epub 2014 Jun 30. PMID 24980612
- [Background] Fan J, McCandliss BD, Sommer T, Raz A, Posner MI. Testing the efficiency and independence of attentional networks. J Cogn Neurosci. 2002 Apr 1;14(3):340-7. doi: 10.1162/089892902317361886. PMID 11970796
- [Background] Goldstone AP, Holland AJ, Butler JV, Whittington JE. Appetite hormones and the transition to hyperphagia in children with Prader-Willi syndrome. Int J Obes (Lond). 2012 Dec;36(12):1564-70. doi: 10.1038/ijo.2011.274. Epub 2012 Jan 24. PMID 22270375
- [Background] Guastella AJ, Einfeld SL, Gray KM, Rinehart NJ, Tonge BJ, Lambert TJ, Hickie IB. Intranasal oxytocin improves emotion recognition for youth with autism spectrum disorders. Biol Psychiatry. 2010 Apr 1;67(7):692-4. doi: 10.1016/j.biopsych.2009.09.020. Epub 2009 Nov 7. PMID 19897177
- [Background] Guastella AJ, Gray KM, Rinehart NJ, Alvares GA, Tonge BJ, Hickie IB, Keating CM, Cacciotti-Saija C, Einfeld SL. The effects of a course of intranasal oxytocin on social behaviors in youth diagnosed with autism spectrum disorders: a randomized controlled trial. J Child Psychol Psychiatry. 2015 Apr;56(4):444-52. doi: 10.1111/jcpp.12305. Epub 2014 Aug 2. PMID 25087908
- [Background] Hall SS, Lightbody AA, McCarthy BE, Parker KJ, Reiss AL. Effects of intranasal oxytocin on social anxiety in males with fragile X syndrome. Psychoneuroendocrinology. 2012 Apr;37(4):509-18. doi: 10.1016/j.psyneuen.2011.07.020. Epub 2011 Aug 20. PMID 21862226
- [Background] Kosfeld M, Heinrichs M, Zak PJ, Fischbacher U, Fehr E. Oxytocin increases trust in humans. Nature. 2005 Jun 2;435(7042):673-6. doi: 10.1038/nature03701. PMID 15931222
- [Background] Lischke A, Gamer M, Berger C, Grossmann A, Hauenstein K, Heinrichs M, Herpertz SC, Domes G. Oxytocin increases amygdala reactivity to threatening scenes in females. Psychoneuroendocrinology. 2012 Sep;37(9):1431-8. doi: 10.1016/j.psyneuen.2012.01.011. Epub 2012 Feb 23. PMID 22365820
- [Background] MacDonald E, Dadds MR, Brennan JL, Williams K, Levy F, Cauchi AJ. A review of safety, side-effects and subjective reactions to intranasal oxytocin in human research. Psychoneuroendocrinology. 2011 Sep;36(8):1114-26. doi: 10.1016/j.psyneuen.2011.02.015. Epub 2011 Mar 23. PMID 21429671
- [Background] Miller JL, Lynn CH, Driscoll DC, Goldstone AP, Gold JA, Kimonis V, Dykens E, Butler MG, Shuster JJ, Driscoll DJ. Nutritional phases in Prader-Willi syndrome. Am J Med Genet A. 2011 May;155A(5):1040-9. doi: 10.1002/ajmg.a.33951. Epub 2011 Apr 4. PMID 21465655
- [Background] Schaller F, Watrin F, Sturny R, Massacrier A, Szepetowski P, Muscatelli F. A single postnatal injection of oxytocin rescues the lethal feeding behaviour in mouse newborns deficient for the imprinted Magel2 gene. Hum Mol Genet. 2010 Dec 15;19(24):4895-905. doi: 10.1093/hmg/ddq424. Epub 2010 Sep 28. PMID 20876615
- [Background] Skokauskas N, Sweeny E, Meehan J, Gallagher L. Mental health problems in children with prader-willi syndrome. J Can Acad Child Adolesc Psychiatry. 2012 Aug;21(3):194-203. PMID 22876265
- [Background] Swaab DF, Purba JS, Hofman MA. Alterations in the hypothalamic paraventricular nucleus and its oxytocin neurons (putative satiety cells) in Prader-Willi syndrome: a study of five cases. J Clin Endocrinol Metab. 1995 Feb;80(2):573-9. doi: 10.1210/jcem.80.2.7852523.
- [Background] Tauber M, Mantoulan C, Copet P, Jauregui J, Demeer G, Diene G, Roge B, Laurier V, Ehlinger V, Arnaud C, Molinas C, Thuilleaux D. Oxytocin may be useful to increase trust in others and decrease disruptive behaviours in patients with Prader-Willi syndrome: a randomised placebo-controlled trial in 24 patients. Orphanet J Rare Dis. 2011 Jun 24;6:47. doi: 10.1186/1750-1172-6-47. PMID 21702900
- [Background] van Lieshout CF, de Meyer RE, Curfs LM, Koot HM, Fryns JP. Problem behaviors and personality of children and adolescents with Prader-Willi syndrome. J Pediatr Psychol. 1998 Apr;23(2):111-20. doi: 10.1093/jpepsy/23.2.111. PMID 9585637
- [Background] Yatawara CJ, Einfeld SL, Hickie IB, Davenport TA, Guastella AJ. The effect of oxytocin nasal spray on social interaction deficits observed in young children with autism: a randomized clinical crossover trial. Mol Psychiatry. 2016 Sep;21(9):1225-31. doi: 10.1038/mp.2015.162. Epub 2015 Oct 27. PMID 26503762